CLINICAL TRIAL: NCT02203357
Title: A Randomized, Opened, Parallel-group Clinical Trial of Hepatitis B Vaccine With Different Dosages and Schedules in Healthy Young Adults
Brief Title: A Randomized,Parallel-group Clinical Trial of Hepatitis B Vaccine With Different Dosages and Schedules in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); Liuzhou City Center for disease control and prevention (Unknown); Shenzhen Kangtai Biological Products Co., LTD (Industry)
Responsible Party: Principal Investigator, Xueen Liu, Dr., Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HepB-2014
Record Dates: First submitted 2014-07-18; First posted 2014-07-29 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B
Keywords: hepatitis B; hepatitis B vaccine; immunogenicity; adults
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

ARMS (3):
- 20μg, 0-1-6 (Active Comparator): 117 young adults were administered with 20μg of hepatitis B vaccine according to the 0-1-6 mon schedule.
  Interventions: Biological: Hepatitis B vaccine
- 60μg, 0-1 (Experimental): 112 young adults were administered with 60μg of hepatitis B vaccine according to the 0-1 mon schedule.
  Interventions: Biological: Hepatitis B vaccine
- 60μg, 0-2 (Experimental): 125 young adults were administered with 60μg of hepatitis B vaccine according to the 0-2 mon schedule.
  Interventions: Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: Hepatitis B vaccine — Hepatitis B vaccine, 60 μg/1ml recombinant hepatitis B vaccine,20 μg/1ml recombinant hepatitis B vaccine, Shenzhen Kangtai Biological Products Co, LTD.

SUMMARY:
The objective of this study is to evaluate the immunogenicity and Anti-HBV antibody persistence of hepatitis B vaccine with different doses and schedules. Hepatitis B vaccine with the regimens of 20μg, 0-1-6 mon and 60μg,0-1 or 0-2 mon will be administered to young adults, and the comparative immunogenicity among the three groups will be measured at 1 mon post-a series vaccination, 1- and 2-year after the first dose of the regimen. Furthermore, the safety of hepatitis B vaccine with different doses and schedules will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 16 and 25 as established by medical history and clinical examination
* Written informed consent will be obtained from each subject before the serum screening of HBV markers
* Seronegative for HBsAg, anti-HBs antibody, anti-HBc antibody
* Have never been immunized with HBV vaccine before

Exclusion Criteria:

* Subject has a medical history of allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Autoimmune disease or immunodeficiency
* Women with pregnant
* Bleeding disorder diagnosed by a doctor
* Chronic diseases: hepatitis, tumor, tuberculosis,et.al
* Any prior administration of immunoglobulins or blood products in the last 3 mon before recruitment
* Subjects had a medical history of serious adverse reactions to vaccines

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 353 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongliao Fang, Dr., Study Director — Guangxi provincial center for desease control and prevention; Hui Zhuang, Dr., Study Director — Peking University Health Science Center
Locations (1):
- Peking University, Beijing, China

REFERENCES:
- [Derived] Wang ZZ, Li MQ, Wang P, Yang ZX, Wei L, Zeng Y, Li YP, Yan L, Liu XE, Zhuang H. Comparative immunogenicity of hepatitis B vaccine with different dosages and schedules in healthy young adults in China. Vaccine. 2016 Feb 17;34(8):1034-9. doi: 10.1016/j.vaccine.2016.01.018. Epub 2016 Jan 19. PMID 26801063

RESULTS

PARTICIPANT FLOW:
Groups:
- 60μg, 0-1: 111 young adults were administered with 60μg of hepatitis B vaccine according to the 0-1 mon schedule.
Period: Overall Study
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Started | 117 | 111 | 125
mon7/2/3 (mon 7 for 0-1-6 group, mon 2 for 0-1 group, mon 3 for 0-2 group) | 114 | 110 | 124
mon12 | 113 | 101 | 122
mon24 | 59 | 45 | 55
Completed | 59 | 45 | 55
Not Completed | 58 | 66 | 70
Not completed — Lost to Follow-up | 58 | 66 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2 | Total
Number analyzed (Participants) | 117 | 111 | 125 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.32 (1.13) | 20.11 (0.94) | 20.18 (1.07) | 20.20 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 42 | 114
  Male | 77 | 79 | 83 | 239
Region of Enrollment [Number; unit: participants]
  China | 117 | 111 | 125 | 353

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of Hepatitis B Vaccine With Different Doses and Schedules in Healthy Young Adults
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA using the Architect i2000SR analyzer (Abbott, Chicago, IL, USA). The accepted protective serum anti-HBs level was ≥10 mIU/ml. Anti-HBs≥10 and < 100 mIU/ml were considered low response, and anti-HBs concentrations ≥100 but < 1000 mIU/ml were middle or moderate response, and hyper or high response was associated with an anti-HBs level ≥1000 mIU/ml.
  The GMCs of anti-HBs antibody will be compared among the three vaccine groups.
Time Frame: one month after a series vaccination of the regimen
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Number analyzed (Participants) | 117 | 111 | 125
mIU/ml | 1847.99 [1417.75 to 2408.8] | 839.27 [507.34 to 1388.35] | 1244.8 [889.61 to 1742.21]
Statistical Analysis 1: Comparison: 20μg, 0-1-6 vs 60μg, 0-1 vs 60μg, 0-2; Test type: Superiority; p < 0.05, ANOVA — The p-value is adjusted for multiple comparisons and the a priori threshold for statistical significance

2. Secondary Outcome: Immunogenicity of Hepatitis B Vaccine With Different Doses and Schedules in Healthy Young Adults
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA using the Architect i2000SR analyzer (Abbott, Chicago, IL, USA). The accepted protective serum anti-HBs level was ≥10 mIU/ml. Anti-HBs≥10 and < 100 mIU/ml were considered low response, and anti-HBs concentrations ≥100 but < 1000 mIU/ml were middle or moderate response, and hyper or high response was associated with an anti-HBs level ≥1000 mIU/ml.
  The GMCs of anti-HBs will be compared among the three vaccine groups.
Time Frame: 1-year after the first dose of the regimens
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Groups:
- 60μg, 0-1: 111young adults were administered with 60μg of hepatitis B vaccine according to the 0-1 mon schedule.
  Hepatitis B vaccine: Hepatitis B vaccine, 60 μg/1ml recombinant hepatitis B vaccine,20 μg/1ml recombinant hepatitis B vaccine, Shenzhen Kangtai Biological Products Co, LTD.
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Number analyzed (Participants) | 113 | 101 | 122
mIU/ml | 1456.63 [1102.78 to 1924.00] | 256.30 [175.70 to 373.85] | 235.15 [172.81 to 319.96]

3. Secondary Outcome: Immunogenicity of Hepatitis B Vaccine With Different Doses and Schedules in Healthy Young Adults
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA using the Architect i2000SR analyzer (Abbott, Chicago, IL, USA). The accepted protective serum anti-HBs level was ≥10 mIU/ml. Anti-HBs≥10 and < 100 mIU/ml were considered low response, and anti-HBs concentrations ≥100 but < 1000 mIU/ml were middle or moderate response, and hyper or high response was associated with an anti-HBs level ≥1000 mIU/ml.
  The GMCs of anti-HBs antibody will be compared among the three vaccine groups. The dynamic changes of seroprotection rates and GMCs of anti-HBs antibody will also be analyzed over the 2 years.
Time Frame: 2-year after the first dose of the regimens
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Number analyzed (Participants) | 59 | 45 | 55
mIU/ml | 427.46 [274.92 to 664.51] | 89.74 [50.43 to 159.70] | 89.80 [56.96 to 141.58]

4. Other Pre Specified Outcome: Safety of HBV Vaccine Determined by Number of Participants With Adverse Events
Description: Participants were monitored for any adverse events occurring within 30 min after each injection for immediate reactions and instructed to measure axillary temperature and record selected injection-site reactions (pain, erythema, induration, swelling, pruritus, cutaneous rash) and systemic reactions (headache, vomiting, asthenia, allergic reaction, fatigue, diarrhea, myalgia, general malaise, etc.) on the day of vaccination and the subsequent 3 days. Adverse reactions were graded or categorized according to the standard guideline for adverse reactions grading in vaccine clinical trials as Grade 1-3.
Time Frame: 0-3 day after the first dose of immunization
Measure: Number; unit: number of participants
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Number analyzed (Participants) | 117 | 111 | 125
number of participants | 2 | 2 | 5

ADVERSE EVENTS:
Arm/Group | 20μg, 0-1-6 | 60μg, 0-1 | 60μg, 0-2
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/111 | 0/125
Other Adverse Events (participants affected / at risk) | 2/117 | 2/111 | 5/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20μg, 0-1-6 (N=117) | 60μg, 0-1 (N=111) | 60μg, 0-2 (N=125)
injection site pain (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No